CLINICAL TRIAL: NCT01111214
Title: Incidence And Serotypes Of Invasive Pneumococcal Disease, After The Introduction Of The Heptavalent Conjugated Vaccine In Greece
Brief Title: Child Pneumococcal Serotype Epidemiology In Greece
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887X1-4434; B1841010
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Pneumococcal Disease
Keywords: Invasive Pneumococcal Disease (IPD); pneumococcal serotypes
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- group 1: Hospitalized children ≤14 years of age with invasive pneumococcal disease
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — There is no intervention. This is a non interventional study.

SUMMARY:
Streptococcus pneumoniae is a major cause of pneumonia, sepsis, bacteremia, and pneumococcal meningitis among infants and children worldwide. The 7-valent conjugate pneumococcal vaccine (Prevenar) has been introduced in the Greek Market in 2004. Additionally, as of 2006 Prevenar has been included in the Greek National Immunization Program.

The effect of the mass vaccination on the incidence of pneumococcal serotypes involved in the occurring invasive pneumococcal disease, is an important factor to consider for the introduction of the 13-valent pneumococcal conjugate vaccine.

DETAILED DESCRIPTION:
open label, one group Purposive sampling of hospitalized children ≤14 years of age with confirmed IPD

ELIGIBILITY:
Inclusion Criteria:

* Children aged 14 years old or less.
* Hospitalized in a participating healthcare facility with an IPD.
* IPD will be confirmed by isolation of S. pneumoniae from a sterile body site.

Exclusion Criteria:

* Children > 14 years of age
* Unconfirmed IPD

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized children in participating centers
Sampling Method: Non-Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The serotype distribution of invasive S. pneumoniae isolates of hospitalized children up to 14 years of age after the introduction of the 7-valent conjugate pneumococcal vaccine | yearly

SECONDARY OUTCOMES:
Serotype distribution of resistant S. pneumoniae isolates | yearly
Serotype distribution of IPD between immunized and non immunized children ≤14 years of age | yearly
Antimicrobial susceptibilities of IPD isolates and rates of resistance to penicillin | yearly

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Greece (9):
  - Agia Sophia Children's Hospital, Athens, Attica
  - University Hospital of Herakleion, Heraklion, Herakleion
  - Venizeleion General Hospital of Herakleion, Heraklion, Herakleion
  - University Hospital of Ioannina, Ioannina, Ioannina
  - Ahepa Hospital Paediatric Outpatient Special Clinic 1st Kyri, Thessaloniki, Thessaloniki
  - Ippokrateion Peripheral Hospital of Thessaloniki, Thessaloniki, Thessaloniki
  - Peripheral Hospital of Trikala, Trikala, Trikala
  - University Hospital of Alexandroupolis, Alexandroupoli
  - University of Thessaly School of Medicine, Larissa

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887X1-4434&StudyName=Child%20Pneumococcal%20Serotype%20Epidemiology%20In%20Greece